CLINICAL TRIAL: NCT03124160
Title: A Multi-center, Single-blind, Randomized Clinical Trial to Compare Two Copper IUDs: Mona Lisa NT Cu380 Mini and ParaGard
Brief Title: Compare Two Copper IUDs: Mona Lisa NT Cu380 Mini and ParaGard
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CCN016
Record Dates: First submitted 2017-02-09; First posted 2017-04-21 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Healthy Women; Female Contraception
Keywords: Healthy Women; Female Contraception; IUD

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mona Lisa® NT Cu380 Mini (Experimental): Mona Lisa® NT Cu380 Mini containing 380mm2 of copper surface inserted into the uterine cavity.
  Interventions: Drug: Mona Lisa® NT Cu380 Mini
- ParaGard® TCu380A (Active Comparator): ParaGard® TCU380A containing 380mm2 of copper surface inserted into the uterine cavity.
  Interventions: Drug: ParaGard® TCu380A

INTERVENTIONS:
Drug: Mona Lisa® NT Cu380 Mini — copper intrauterine device
  Other Names: NT380-Mini, NTCu380-Mini
  Arms: Mona Lisa® NT Cu380 Mini
Drug: ParaGard® TCu380A — copper intrauterine device
  Other Names: T380
  Arms: ParaGard® TCu380A

SUMMARY:
This will be a multi-site, participant-blinded, randomized clinical trial. The investigators will randomize 1000 eligible participants in a 4:1 ratio to two different copper IUDs: 800 to Mona Lisa NT Cu380 Mini and 200 to ParaGard.

DETAILED DESCRIPTION:
The total duration of the study for each participant is expected to be approximately 39 months: including screening and enrollment (up to 30 days to meet enrollment criteria), 37 months of participation, and a post-removal follow up telephone call 17 days post-removal. After enrollment, subject visits occur at 6 weeks, 3 months, 6 months, 12 months, 24 months, with telephone calls at 9, 18, and 30 months and seen again at 37 months for their final visit. Subjects will use a home pregnancy test 17 days post-removal of the IUD or Exit Visit procedures, whichever occurs first, and called by the site for the result and for safety follow-up.

Subject recruitment is expected to begin Q2 (in the second quarter of) 2017 and is planned to continue through Q2 2018. However, if the enrollment rate declines, the enrollment period may be extended beyond this date. If this enrollment timeline is met, all subjects should finish active treatment by approximately the end of Q2 2021. The total duration of the study will be approximately 48 months for each study site including pre- and post- trial activities. The end of the study will occur when the last subject to be enrolled has completed her post-removal pregnancy test telephone call.

Total duration of the project is expected to be five years. Preliminary results of the study are expected to be available Q4 of 2019 based on the current study plan.

ELIGIBILITY:
Inclusion Criteria:

* 16-40 years

  o 16 and 17 year olds, where permissible by state regulations and local Institutional Review Board (IRB) approval
* Sexually active, anticipating at least one act of vaginal intercourse per menstrual cycle with a male partner and at risk for pregnancy
* seeking contraception, and willing to use the study IUD as the only contraception method
* willing to be randomized to one of the two copper IUDs
* has an intact uterus and at least one ovary
* has a history of regular menstrual cycles; defined as occurring every 21-35 days when not using hormones, and with a variation of typical cycle length of no more than 5 days
* able and willing to provide written informed consent
* agrees to follow all study requirements
* not currently pregnant or at risk for luteal phase pregnancy based on history of unprotected intercourse

Exclusion Criteria:

* abnormal Pap requiring treatment after enrollment
* known human immunodeficiency virus / acquired immunodeficiency syndrome (HIV/AIDS) infection
* intending to become pregnant in the 37 months after enrollment
* known infertility
* history of allergy or sensitivity to copper
* previous tubal sterilization
* has received an injectable contraceptive in the last 9 months and has not resumed regular menstrual cycles (as evidenced by 2 spontaneous menses)
* within 30 days of administration of mifepristone and/or misoprostol for medical abortion or for miscarriage management
* within 30 days of first, second, or third trimester abortion or miscarriage (note: potential abortion/miscarriage participants can be screened and return after 30 days for randomization and IUD insertion)
* within 30 days of delivery (for parous population)
* breastfeeding or recently breastfeeding women unless two consecutive normal menstrual periods have occurred after delivery and prior to enrollment.
* wants to use a copper IUD for emergency contraception
* has previously participated in the study
* participated in another clinical trial involving an investigational product within the last 30 days (before screening) or planning to participate in another clinical trial involving an intervention or treatment during this study
* not living in the catchment area of the study site or planning to move from the area within the year (unless known to be moving to the catchment area of another study site)
* known or suspected current alcohol or drug abuse
* planning to undergo major surgery during study participation
* current need for use of exogenous hormones or therapeutic anticoagulants (Note: subjects who start a therapeutic anticoagulant after enrolment will be allowed to continue in the study.)
* at high risk for sexually-transmitted infections or pelvic infection
* anticipated need for regular condom use (refer to Section 8.1).
* has any condition (social or medical) which in the opinion of the Investigator would make study participation unsafe or complicate data interpretation
* Reported medical contraindications (Medical Eligibility Criteria category 3 or 4)14 to copper IUDs, including:

  * suspicious unexplained vaginal bleeding
  * known cervical cancer
  * known endometrial cancer
  * known Wilson's disease
  * Confirmed gestational trophoblastic disease with persistently elevated beta-hCG levels or malignant disease, with evidence or suspicion of intrauterine disease
  * anatomic abnormalities with distorted uterine cavity
  * current pelvic inflammatory disease (PID)
  * pelvic tuberculosis
  * immediately post-septic abortion or puerperal sepsis
  * current known purulent cervicitis or chlamydial infection or gonorrhea; Note: to enroll, there must be no obvious signs of infection at the time of enrollment based on pelvic exam. If lab results come back for positive infection after enrollment, treatment should be provided but the IUD can be left in place.
  * complicated solid organ transplantation
  * systemic lupus erythematosus with severe thrombocytopenia

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1105 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Blithe, Study Director — National Institute of Child Health & Human Development (NICHD); David Hubacher, Study Director — FHI 360
Locations (16):
- United States (16):
  - Essential Access Health, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Denver, Colorado
  - University of Hawaii, Honolulu, Hawaii
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Medical Center Corporation, Boston, Massachusetts
  - Planned Parenthood League of Massachusetts, Boston, Massachusetts
  - Planned Parenthood of New York, New York, New York
  - Columbia University, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sivin I, Stern J. Long-acting, more effective copper T IUDs: a summary of U.S. experience, 1970-75. Stud Fam Plann. 1979 Oct;10(10):263-81. No abstract available. PMID 516121
- [Background] Sivin I, Tatum HJ. Four years of experience with the TCu 380A intrauterine contraceptive device. Fertil Steril. 1981 Aug;36(2):159-63. PMID 7262334
- [Background] Sivin I, Stern J, Coutinho E, Mattos CE, el Mahgoub S, Diaz S, Pavez M, Alvarez F, Brache V, Thevenin F, et al. Prolonged intrauterine contraception: a seven-year randomized study of the levonorgestrel 20 mcg/day (LNg 20) and the Copper T380 Ag IUDS. Contraception. 1991 Nov;44(5):473-80. doi: 10.1016/0010-7824(91)90149-a. PMID 1797462
- [Background] The TCu380A, TCu220C, multiload 250 and Nova T IUDS at 3,5 and 7 years of use--results from three randomized multicentre trials. World Health Organization. Special Programme of Research, Development and Research Training in Human Reproduction: Task Force on the Safety and Efficacy of Fertility Regulating Methods. Contraception. 1990 Aug;42(2):141-58. PMID 2085966
- [Background] Hubacher D. Copper intrauterine device use by nulliparous women: review of side effects. Contraception. 2007 Jun;75(6 Suppl):S8-11. doi: 10.1016/j.contraception.2006.12.005. Epub 2007 Feb 20. PMID 17531622
- [Background] Abraham M, Zhao Q, Peipert JF. Young Age, Nulliparity, and Continuation of Long-Acting Reversible Contraceptive Methods. Obstet Gynecol. 2015 Oct;126(4):823-829. doi: 10.1097/AOG.0000000000001036. PMID 26348177
- [Background] Benacerraf BR, Shipp TD, Lyons JG, Bromley B. Width of the normal uterine cavity in premenopausal women and effect of parity. Obstet Gynecol. 2010 Aug;116(2 Pt 1):305-310. doi: 10.1097/AOG.0b013e3181e6cc10. PMID 20664389
- [Background] Koch P, Reinhardt P, Soyka E. Intrauterine contraception using the Copper Mini-Gravigard 7 IUD: summary of 328 case histories. Contracept Deliv Syst. 1981 Apr;2(1):171-6. PMID 12336868
- [Background] Petersen KR, Brooks L, Jacobsen N, Skoby SO. Clinical performance of intrauterine devices in nulligravidae: is the length of the endometrial cavity of significance? Acta Eur Fertil. 1991 Jul-Aug;22(4):225-8. PMID 1844327
- [Background] Otero-Flores JB, Guerrero-Carreno FJ, Vazquez-Estrada LA. A comparative randomized study of three different IUDs in nulliparous Mexican women. Contraception. 2003 Apr;67(4):273-6. doi: 10.1016/s0010-7824(02)00519-x. PMID 12684147
- [Background] Ott MA, Sucato GS; Committee on Adolescence. Contraception for adolescents. Pediatrics. 2014 Oct;134(4):e1257-81. doi: 10.1542/peds.2014-2300. PMID 25266435
- [Background] Committee on Adolescent Health Care Long-Acting Reversible Contraception Working Group, The American College of Obstetricians and Gynecologists. Committee opinion no. 539: adolescents and long-acting reversible contraception: implants and intrauterine devices. Obstet Gynecol. 2012 Oct;120(4):983-8. doi: 10.1097/AOG.0b013e3182723b7d. PMID 22996129
- [Background] Curtis KM, Tepper NK, Jatlaoui TC, Berry-Bibee E, Horton LG, Zapata LB, Simmons KB, Pagano HP, Jamieson DJ, Whiteman MK. U.S. Medical Eligibility Criteria for Contraceptive Use, 2016. MMWR Recomm Rep. 2016 Jul 29;65(3):1-103. doi: 10.15585/mmwr.rr6503a1. PMID 27467196
- [Background] Heinemann K, Reed S, Moehner S, Minh TD. Risk of uterine perforation with levonorgestrel-releasing and copper intrauterine devices in the European Active Surveillance Study on Intrauterine Devices. Contraception. 2015 Apr;91(4):274-9. doi: 10.1016/j.contraception.2015.01.007. Epub 2015 Jan 16. PMID 25601352
- [Background] Farley TM, Rosenberg MJ, Rowe PJ, Chen JH, Meirik O. Intrauterine devices and pelvic inflammatory disease: an international perspective. Lancet. 1992 Mar 28;339(8796):785-8. doi: 10.1016/0140-6736(92)91904-m. PMID 1347812
- [Derived] Schreiber CA, Nanda K, Hubacher D, Turok DK, Jensen JT, Creinin MD, White KO, Dayananda I, Teal SB, Chen PL, Chen BA, Goldberg AB, Kerns JL, Dart C, Nelson AL, Thomas MA, Archer DF, Brown JE, Castano PM, Burke AE, Kaneshiro B, Blithe DL. Contraceptive Efficacy and Comparative Side Effects of a Mini Copper Intrauterine Device. NEJM Evid. 2025 Aug;4(8):EVIDoa2400480. doi: 10.1056/EVIDoa2400480. Epub 2025 Jul 22. PMID 40693846
- [Derived] Hubacher D, Schreiber CA, Turok DK, Jensen JT, Creinin MD, Nanda K, White KO, Dayananda I, Teal SB, Chen PL, Chen BA, Goldberg AB, Kerns JL, Dart C, Nelson AL, Thomas MA, Archer DF, Brown JE, Castano PM, Burke AE, Kaneshiro B, Blithe DL. Continuation rates of two different-sized copper intrauterine devices among nulliparous women: Interim 12-month results of a single-blind, randomised, multicentre trial. EClinicalMedicine. 2022 Jul 16;51:101554. doi: 10.1016/j.eclinm.2022.101554. eCollection 2022 Sep. PMID 35865736
- See also: NDA for Paragard (TCu380A) — http://www.accessdata.fda.gov/drugsatfda_docs/label/2013/018680s066lbl.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Mona Lisa® NT Cu380 Mini: Mona Lisa® NT Cu380 Mini containing 380mm2 of copper surface inserted into the uterine cavity.
  Mona Lisa® NT Cu380 Mini: Mona Lisa® NT Cu380 Mini
- ParaGard® TCu380A: ParaGard® TCU380A containing 380mm2 of copper surface inserted into the uterine cavity.
  ParaGard® TCu380A: ParaGard® TCu380A
Period: Overall Study
Arm/Group | Mona Lisa® NT Cu380 Mini | ParaGard® TCu380A
Started | 887 | 218
Completed | 426 | 91
Not Completed | 461 | 127

BASELINE CHARACTERISTICS:
Population: Females aged 17-40 interested in using a contraceptive method
Groups:
- Total: Total of all reporting groups
Arm/Group | Mona Lisa® NT Cu380 Mini | ParaGard® TCu380A | Total
Number analyzed (Participants) | 887 | 218 | 1105
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline count of participants
  years | 26.3 (5.23) | 26.3 (4.96) | 26.3 (5.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 887 | 218 | 1105
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 117 | 31 | 148
  Not Hispanic or Latino | 765 | 187 | 952
  Unknown or Not Reported | 5 | 0 | 5
Number of Participants [Count of Participants; unit: Participants] | 887 | 218 | 1105

OUTCOME MEASURES:

1. Primary Outcome: Pregnancy Rate of Mona Lisa Copper IUD Over 3 Years
Description: Pearl Index is a measure of contraceptive efficacy used by the FDA that summarizes number of method failures per 100 person years
Time Frame: 3 years
Population: includes only participants with an evaluable cycle for estimating efficacy
Measure: Number (95% Confidence Interval); unit: Pearl Index = Num preg per 100 person yr
Groups:
- Mona Lisa NT Cu380 Mini Participants <36 Years of Age: This is the FDA definition and uses evaluable cycles in the denominator and failures in the numerator, summarized in failures per 100 person years.
Arm/Group | Mona Lisa NT Cu380 Mini Participants <36 Years of Age
Number analyzed (Participants) | 804
Pearl Index = Num preg per 100 person yr | 1.86 [1.20 to 2.74]

2. Secondary Outcome: IUD Continuation
Description: IUD continuation at 36-months by product
Time Frame: 3 years
Population: Participants with successful IUD insertion
Measure: Count of Participants; unit: Participants
Arm/Group | Mona Lisa® NT Cu380 Mini | ParaGard® TCu380A
Number analyzed (Participants) | 875 | 213
Participants | 426 | 91

3. Secondary Outcome: Failed IUD Insertion
Description: Failed IUD insertion as measured by inability to place the IUD correctly
Time Frame: Immediate after IUD insertion attempt
Population: Treated population: uterus was successfully sounded and IUD insertion attempt was made
Measure: Number; unit: participants
Arm/Group | Mona Lisa® NT Cu380 Mini | ParaGard® TCu380A
Number analyzed (Participants) | 876 | 214
participants | 1 | 1

4. Secondary Outcome: Uterine Perforation
Description: Uterine perforation as measured by ultrasound
Time Frame: 3 years
Population: User population
Measure: Count of Participants; unit: Participants
Arm/Group | Mona Lisa® NT Cu380 Mini | ParaGard® TCu380A
Number analyzed (Participants) | 875 | 213
Participants | 1 | 0

5. Secondary Outcome: IUD Expulsion (Complete and Partial)
Description: When the IUD is expelled from the uterus, either completely or partially.
Time Frame: 3 years
Population: user population
Measure: Count of Participants; unit: Participants
Arm/Group | Mona Lisa® NT Cu380 Mini | ParaGard® TCu380A
Number analyzed (Participants) | 875 | 213
Participants | 66 | 22

6. Secondary Outcome: Vaginal Bleeding Patterns
Description: Proportion of cycles with heavy bleeding (more than 4 sanitary products in a day)
Time Frame: 1 year
Population: User population with evaluable cycles
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: Number of 28-day cycles
Arm/Group | Mona Lisa® NT Cu380 Mini | ParaGard® TCu380A
Number analyzed (Participants) | 875 | 213
Number analyzed (Number of 28-day cycles) | 9292 | 2185
percent | 54.4 [53.43 to 55.46] | 55.7 [53.54 to 57.75]

7. Secondary Outcome: Pelvic Pain as Measured in the Subject Diary
Description: Percent of cycles with any pelvic pain will be calculated using all available cycles
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percent
Units Other Than Participants: Number of 28-day cycles
Arm/Group | Mona Lisa® NT Cu380 Mini | ParaGard® TCu380A
Number analyzed (Participants) | 875 | 213
Number analyzed (Number of 28-day cycles) | 9292 | 2185
percent | 72.3 [71.3 to 73.2] | 72.3 [70.4 to 74.1]

8. Secondary Outcome: Dysmenorrhea
Description: Number of participants who experienced any dysmenorrhea during the trial
Time Frame: 3 years
Population: User population
Measure: Count of Participants; unit: Participants
Arm/Group | Mona Lisa® NT Cu380 Mini | ParaGard® TCu380A
Number analyzed (Participants) | 875 | 213
Participants | 396 | 100

9. Secondary Outcome: Pain With and Shortly After Insertion as Recorded by Study Subjects
Description: Pain level on scale of 0=no pain to 10=worst imaginable pain as displayed on a paper form for study subject to indicate their level of pain
Time Frame: Pain level 10 minutes after IUD insertion
Population: User population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mona Lisa® NT Cu380 Mini | ParaGard® TCu380A
Number analyzed (Participants) | 875 | 213
units on a scale | 1.8 (1.92) | 2.1 (1.83)

10. Secondary Outcome: Ease of IUD Insertion as Recorded by the Investigator
Description: Investigator to assess ease of IUD insertion (easy, somewhat easy, somewhat hard or hard)
Time Frame: Right after IUD insertion
Measure: Count of Participants; unit: Participants
Arm/Group | Mona Lisa® NT Cu380 Mini | ParaGard® TCu380A
Number analyzed (Participants) | 875 | 213
Participants
  Easy | 694 | 161
  Somewhat easy | 132 | 43
  Somewhat hard | 41 | 6
  Hard | 8 | 3

11. Secondary Outcome: Overall Product Satisfaction as Measured by Acceptability Questions Asked of Subjects
Description: Overall product satisfaction level at exit visit (highly satisfied, satisfied, dissatisfied, highly dissatisfied)
Time Frame: 3 years
Population: User population
Measure: Count of Participants; unit: Participants
Arm/Group | Mona Lisa® NT Cu380 Mini | ParaGard® TCu380A
Number analyzed (Participants) | 761 | 194
Participants
  Highly satisfied | 364 | 92
  Satisfied | 248 | 49
  Dissatisfied | 118 | 43
  Highly dissatisfied | 31 | 10

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Mona Lisa® NT Cu380 Mini | ParaGard® TCu380A
All-Cause Mortality (participants affected / at risk) | 0/887 | 0/218
Serious Adverse Events (participants affected / at risk) | 32/887 | 3/218
Other Adverse Events (participants affected / at risk) | 742/875 | 183/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mona Lisa® NT Cu380 Mini (N=887) | ParaGard® TCu380A (N=218)
appendicitis (Infections and infestations) | 8 (8) | 0 (0)
pyelonephritis (Infections and infestations) | 4 (4) | 0 (0)
infected bite (Infections and infestations) | 1 (1) | 0 (0)
tubo-ovarian abscess (Infections and infestations) | 1 (1) | 0 (0)
enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
suicidal ideation (Psychiatric disorders) | 2 (2) | 0 (0)
suicidal attempt (Psychiatric disorders) | 2 (2) | 0 (0)
dependence (Psychiatric disorders) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 1 (1) | 0 (0)
limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
open fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
uterine perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0)
ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
premature delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
appendicectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
thyroid nodule removal (Surgical and medical procedures) | 1 (1) | 0 (0)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ovarian mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
pre-eclampsia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mona Lisa® NT Cu380 Mini (N=875) | ParaGard® TCu380A (N=213)
dysmenorrhoea (Reproductive system and breast disorders) | 390 (494) | 100 (123)
menorrhagia (Reproductive system and breast disorders) | 315 (477) | 82 (112)
metrorrhagia (Reproductive system and breast disorders) | 250 (334) | 54 (61)
pelvic pain (Reproductive system and breast disorders) | 186 (246) | 46 (48)
uterine spasm (Reproductive system and breast disorders) | 71 (101) | 22 (34)
dyspareunia (Reproductive system and breast disorders) | 61 (64) | 8 (8)
procedural pain (Injury, poisoning and procedural complications) | 511 (574) | 135 (150)
abdominal pain (Gastrointestinal disorders) | 61 (80) | 16 (23)
bacterial vaginosis (Infections and infestations) | 48 (60) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT03124160/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT03124160/SAP_001.pdf
  • Informed Consent Form (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT03124160/ICF_002.pdf